CLINICAL TRIAL: NCT04883866
Title: Impact of Telephone Breastfeeding Support on Breastfeeding Outcomes for Mothers With Premature Babies: Randomized Controlled Study
Brief Title: Phone Breastfeeding Support for Premature Babies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ezgi Boz, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KAEK- 118
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Preterm Birth; Breastfeeding
Keywords: Telephone based support,
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Intervention Model Description: This is a pretest-posttest designed randomized controlled trial using the stratified block randomization method.
Who Masked: Participant, Outcomes Assessor
Masking Description: At the time of discharge, the participants will not know that they are in the intervention and control group. Participants will be blinded. In the evaluation of the data, the groups will not be coded as intervention and control groups, they will be coded as group A and group B, and their analysis will be evaluated and reported by an independent statistician. In addition, the statistician will be blind.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Sending breastfeeding guidelines for premature babies to phones after the discharge procedure is completed.and implementing a "Telephone Breastfeeding Support Program".
  Interventions: Behavioral: Telephone Breastfeeding Support Program; Behavioral: Sending a breastfeeding guide for premature babies to the phone of mothers in addition to the routine discharge procedure
- Control Group (Experimental): Sending breastfeeding guidelines for premature babies to phones after the discharge procedure is completed.
  Interventions: Behavioral: Sending a breastfeeding guide for premature babies to the phone of mothers in addition to the routine discharge procedure

INTERVENTIONS:
Behavioral: Telephone Breastfeeding Support Program — On the 3rd day after discharge, a reminder messages will be sent to the mothers in the inter vention group. Throughout the program, 21 reminder messages will be sent to mothers in the first month after discharge to support the mother and encourage breast milk via a messaging application (whatsapp, bip, telegram, etc.). In addition, a total of seven phone calls, once a week in the first month after discharge and once a month in the eighth, twelfth and sixteenth weeks, will be made to check personalized information about individual breastfeeding questions of mothers.
  Arms: Intervention Group
Behavioral: Sending a breastfeeding guide for premature babies to the phone of mothers in addition to the routine discharge procedure — In addition to the routine discharge procedure, a breastfeeding guide for premature babies will be sent to the mothers' phone.

SUMMARY:
It was observed that premature babies had the risk of insufficient milk intake and a lower rate of breastfeeding compared to term babies. Various problems may occur at home, especially after breastfeeding training in the hospital. After discharge, support and counseling should be provided to eliminate problems that may stop breastfeeding or to prevent events that may prevent breastfeeding. The aim of this study is to examine the effect of "Telephone Breastfeeding Support" given to mothers of premature babies discharged from the neonatal intensive care unit on breastfeeding results.

DETAILED DESCRIPTION:
The study was planned as a randomized, parallel two-group, controlled experimental design. This research will be conducted between June 2021 and June 2022 with premature baby mothers. The sample of the study will be mothers (n = 62) of premature babies discharged from Antalya Training and Research Hospital Neonatal Intensive Care Unit. The discharge routine procedures of all mothers participating in the study will be completed and a breastfeeding guide prepared for premature babies will be sent to the phone. On the 3rd day after discharge, a reminder message will be sent to support the mother in the intervention group (n = 31) and to encourage breast milk. Throughout the program, 21 messages will be sent to the mothers in the first month after discharge, via the messaging application (whatsapp, bip, telegram, etc.) In addition, seven phone calls will be made once a week in the first month after discharge, and once a month in the eighth, twelfth and sixteenth weeks. Data will be collected by Mother-Baby Introductory Information Form, Breastfeeding Self-Efficacy Scale (short form) (BSES), Infant Feeding Attitude Scale (IIFAS) and Breastfeeding Time Assessment Form. The pre-test will be taken with the Mother-Baby Descriptive Information Form, BSES and IIFAS during the discharge routine procedures, and the post-test will be taken with the BSES, IIFAS and Breastfeeding Time Assessment Form when the baby is six months old. Ethics Committee and Institutional Permission was obtained for the study. In addition, written consent will be obtained from the participants. Statistical analysis will be done using SPSS 23.0 and significance will be evaluated at p <0.05. Support will be received in the analysis phase of the Statistical Information Unit of Akdeniz University. It is anticipated that new information from research data will improve breastfeeding results of premature babies and guide new research.

ELIGIBILITY:
Inclusion Criteria:

* Whose baby was born between 34 weeks + 0 days and 36 weeks + 6 days (late preterms),
* Does not have severe congenital anomalies in her baby (according to hospital records),
* Breastfeeding her baby,
* Reading and writing,
* Can speak and understand Turkish,
* Mothers who agreed to participate in the study,
* Mothers having a smartphone.

Exclusion Criteria:

* Mothers with previous experience of breastfeeding a premature baby,
* Plural baby,
* Mother's breastfeeding disability (according to hospital records).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy Scale (short form) | 0-6 months (During discharge routine procedures and when the baby is six months old)
  The scale, which is valid and reliable in our country by Aluş Tokat, Okun and Dennis (2010), consists of 14 items and is a Likert type scale rated between 1 and 5. The minimum score that can be retrieved from the scale is 14 and the maximum is 70. As the score rises, high breastfeeding is an indicator of self-sufficiency.
Infant Feeding Attitude Scale | 0-6 months (During discharge routine procedures and when the baby is six months old)
  The scale was developed to evaluate women's attitudes towards breastfeeding and to predict breastfeeding duration as well as the choice of baby feeding method. The scale consists of 5-point Likert type and 17 items. The total attitude score ranges from 17 (showing a positive attitude to bottle feeding) to 85 (reflecting a positive attitude towards breastfeeding). The higher the score on the scale, the higher it indicates the higher breastfeeding attitude.
3. Breastfeeding Time Evaluation Form Breastfeeding Time Evaluation Form Breastfeeding Time Evaluation Form | When the baby is six months old
  Prepared by researcher to find out breastfeeding status when babies are 6 months old.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Akcan, PhD, Study Director — +905334436659
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No